CLINICAL TRIAL: NCT00386620
Title: Spousal Relationships and Pain in Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2003-0595; W81XWH-04-1-0425 (Other: Department of Defense Breast Cancer Research Program)
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cancer Control; Spousal Relationships; Questionnaire; Interview; Pain
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey + ED: Part 1: Survey + Electronic Diaries (ED)
  Part 2: 3 Month, 6 Month Survey + ED
  Interventions: Behavioral: Questionnaire; Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaire — 45 minute survey about health, pain and relationships
Behavioral: Interview — Feedback on use of handheld computer electronic diaries (ED).

SUMMARY:
Ecological Momentary Assessment (EMA) refers to the collection of repeated measurements of phenomena as they occur in naturalistic settings using hand-held computers. By providing an EMA of psychosocial variables that influence patient pain and pain behaviors, this study seeks to characterize the pain experience in metastatic breast cancer from both patients' and spouses' perspectives.

This study consists of two parts. Part 1 involves developing and pilot testing a hand-held computer program designed to assess antecedents, behaviors, and consequences of patient pain, as well as spouse response to pain. Five couples will complete a baseline survey and carry the hand-held computer for two weeks. They will be interviewed for feedback to refine the program. Part 2 is a longitudinal assessment of the psychological and relationship functioning of metastatic breast cancer patients and their spouses. The Optional Procedure for Part 2 involves using electronic diaries (EDs) to measure the cancer pain experience for patients with metastatic breast cancer and their spouses.

The specific aims of this study are to: (1) To examine patient pain, spouse response to patient pain, and patient behaviors in response to pain over the course of 6 months in couples facing metastatic breast cancer, (2) test the biopsychosocial model of chronic pain in breast cancer; expanding it to include the influence of patient psychological functioning, spouse psychological functioning, and relationship functioning, on patient pain, spouse behaviors, and patient behaviors in response to pain, (3) use ecological momentary assessment to characterize patient pain, spouse response to patient pain, and patient behaviors in response to pain.

DETAILED DESCRIPTION:
Part 1:

Women with metastatic breast cancer will be asked to take part in the study. Project staff will review patients' medical records to determine their eligibility for the study. Eligible patients will be approached by a project staff member when they begin treatment for metastatic disease.

By agreeing to participate, you are agreeing to allow the study staff to contact your spouse. Spouses who are not present at the time patients are consented will not be asked to participate. Interested patients may still participate in this study even if their spouse is unwilling or unable to participate.

A project staff member will show participants how to use hand-held computers. Learning to use the computers does not require previous computer experience. Participants will take the computers home and, when signaled by the computer, answer a brief series of questions about how they are feeling physically and emotionally at that particular moment.

Participants will be prompted to answer questions 6 times a day, for 14 days after starting treatment. It should take about 2 minutes to answer the questions each time.

Upon completion, participants will be interviewed separately in person or on the telephone for feedback about using the computer. The interview should take about 30 minutes.

At the time participants are consented, they will also be asked to complete several questionnaires about their health, pain, and their relationship. It will take about 45 minutes to complete all of the questionnaires. Participants may complete the questionnaires while waiting for their clinic appointments, or they may take the questionnaires home, complete them, and return them in a pre-stamped envelope.

A project staff member will review patients' medical records to collect medical information relevant to this study.

All answers given by participants will be kept private.

This is an investigational study. A total of 5 patients and 5 spouses will be asked to participate. All we be enrolled at M. D. Anderson.

Part 2:

Women with metastatic breast cancer will be asked to take part in the study. Project staff will review patients' medical records to determine their eligibility for the study. Eligible patients will be approached by a project staff member when they begin treatment for metastatic disease.

By agreeing to participate, you are agreeing to allow the study staff to contact your spouse. Spouses who are not present at the time patients are consented will be contacted by phone, to find out if they are interested in participating in this study.

Patients and spouses who are interested in participating will be asked to complete several questionnaires about their health, pain, and their relationship. It will take about 45 minutes to complete all of the questionnaires. Participants in this study may complete the questionnaires while waiting for their clinic appointments, or they may take the questionnaires home, complete them, and return them in a pre-stamped envelope.

Both patients and their spouses will be asked to complete the same questionnaires 3 months after completing the first questionnaire, and then again 3 months later. Any patient whose spouse does not wish to participate will not be asked to complete these additional questionnaires.

Attempts will be made to give these questionnaires during routine clinic appointments so that the questionnaires can be completed while in the waiting room. If appointments do not occur at the same time as the questionnaires are scheduled to be completed or clinic time does not permit, patients and spouses will be mailed the questionnaire packets and asked to return them in self-addressed stamped envelopes.

A project staff member will review patients' medical records to collect medical information relevant to this study.

All answers given by participants will be kept private.

This is an investigational study. Up to 622 individuals (311 patients and 311 spouses) will be asked to participate in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. For Patients: Being a female patient diagnosed with metastatic breast cancer.
2. For Patients: Initiating treatment for metastatic breast cancer
3. For Patients: Having and ECOG Performance Status Score of 2 or less
4. For Spouses: Being the male spouse or significant other of a female patient diagnosed with metastatic breast cancer
5. For Spouses: Having the patient's consent to be contacted
6. For Patients and Spouses: Having the ability to read and speak English well enough to understand the consent form and complete the questionnaires
7. For Patients and Spouses: Being able to provide informed consent

Exclusion Criteria:

1. For Patients and Spouses: Not being able to provide informed consent.
2. For Patients: Rating average pain as 0 on the BPI

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women diagnosed with metastatic breast cancer and their male spouse or significant other
Sampling Method: Non-Probability Sample
Enrollment: 548 (Actual)
Dates: Start 2004-10; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Longitudinal assessment of the psychological and relationship functioning of metastatic breast cancer patients and their spouses. | 6 Months

SECONDARY OUTCOMES:
Pilot of hand-held computers at home for metastatic breast cancer patient and spouses to answer questions about pain and other symptoms. | 14 Days (Survey Response + 30 Minute Interview)

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Badr, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org